CLINICAL TRIAL: NCT04245449
Title: A Novel Therapy + E-learning Self-management Program for Stroke Survivors
Brief Title: E-learning+ Rehab Therapy
Acronym: TEAACH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19 and loss of funding
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Michelle Woodbury, Associate Professor, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00081749; P20GM109040-06 (NIH)
Record Dates: First submitted 2020-01-21; First posted 2020-01-29 (Actual); Results first posted 2023-01-26 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- e learning+therapy (TEAACH) (Experimental): TEAACH-Training to Empower Activity-dependent plasticity-based Arm-use habits in the Community and at Home
  Interventions: Behavioral: TEAACH

INTERVENTIONS:
Behavioral: TEAACH — TEAACH e-learning: 3-months of online educational modules include neuroscience education (based on an effective pain educational model37) to improve patient self-efficacy, and strategy-training38 to improve patients' problem-solving abilities for at-home arm use. The course is live on the MUSC MoodleCE platform.
  TEAACH in-clinic therapy: 24 in-clinic sessions; 3 times/week for 4 weeks (month 1), 2 times/week for 4 weeks (month 2) and 1 time/week for 4 weeks (month 3) with 200 movement repetitions per session. In our RCTs, this therapy dose required ~1.0-1.5 hours/session. A critical element of TEAACH is the focus on linking in-clinic therapy to out-of-clinic real world paretic arm use via MoodleCE Learning Activities.

SUMMARY:
Stroke survivors with arm paresis because of stroke use their "good" arm for daily activities, but in doing so may be self-limiting their own recovery of the "bad" arm. Traditional models of stroke rehabilitation fail to fully engage the survivor and care partner(s) in actively planning post-discharge habits that improve their capacity to live well over their entire lives. This study will test a cutting-edge in-person therapy + online training program designed to progressively transfer the responsibility of driving post-stroke recovery from the therapist to the survivor.

ELIGIBILITY:
Inclusion Criteria:

* paresis of one arm/hand because of ischemic or hemorrhagic stroke >2 mo. and <3 yrs prior
* moderate arm impairment defined as a baseline Fugl-Meyer Assessment of the Upper Extremity score of at least 32±2 points but no more than 47±2 points (out of 60 points)
* Montreal Cognitive Assessment score ≥22
* ability to read English
* ability to communicate as per the therapists' judgement at baseline testing
* 21-90 years of age
* wi-fi connection in the home and either a computer, smartphone or tablet.

Exclusion criteria:

* lesion or injury to brainstem or cerebellum
* other neurological disease that may impair motor or learning skills (e.g., Parkinson's Disease);
* pain interfering with reaching
* uncorrected vision making it difficult to read information on a computer, tablet or phone.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Woodbury, PT, PhD, Principal Investigator — Medical University of SC
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were enrolled however the study is designed so that cohorts start together. Study procedures did not start until a group of subjects were enrolled. Due to Covid shutting the study down study procedures did not start.
Groups:
- e Learning+Therapy (TEAACH): TEAACH-Training to Empower Activity-dependent plasticity-based Arm-use habits in the Community and at Home
  TEAACH: TEAACH e-learning: 3-months of online educational modules include neuroscience education (based on an effective pain educational model37) to improve patient self-efficacy, and strategy-training38 to improve patients' problem-solving abilities for at-home arm use. The course is live on the MUSC MoodleCE platform.
  TEAACH in-clinic therapy: 24 in-clinic sessions; 3 times/week for 4 weeks (month 1), 2 times/week for 4 weeks (month 2) and 1 time/week for 4 weeks (month 3) with 200 movement repetitions per session. In our RCTs, this therapy dose required ~1.0-1.5 hours/session. A critical element of TEAACH is the focus on linking in-clinic therapy to out-of-clinic real world paretic arm use via MoodleCE Learning Activities.
Period: Overall Study
Arm/Group | e Learning+Therapy (TEAACH)
Started | 7
Completed | 0
Not Completed | 7
Not completed — COVID shutdown | 7

BASELINE CHARACTERISTICS:
Arm/Group | e Learning+Therapy (TEAACH)
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Health Literacy From Baseline to 3 Months
Description: Health Literacy will be assessed via a standardize 18-item test designed to assess an adult's ability to read and understand common medical terms. Minimum = 0, Maximum = 18. Higher scores indicate greater health literacy.
Time Frame: Baseline Visit and 3 months
Population: Although the first subject was enrolled in August 2019, the Project was designed so that a cohort started together. In other words, the study team could not start study procedures until we had a group of subjects enrolled. Hence, although the first participant was enrolled in August, the study team was not able to start the study, because of the covid shut down in March prior to beginning the group related study procedures.
Arm/Group | e Learning+Therapy (TEAACH)
Number analyzed (Participants) | 0

2. Primary Outcome: Change in Self Management Skills From Baseline to 3 Months
Description: Participants' ability to manage their chronic condition (their stroke) will be assessed qualitatively using interview questions. Participants' narratives will be analyzed and reported as a description of how their own skills have changed.
Time Frame: Baseline and 3 months
Population: as for outcome 1
Arm/Group | e Learning+Therapy (TEAACH)
Number analyzed (Participants) | 0

3. Secondary Outcome: Change in Self-Efficacy for Managing Daily Activities From Baseline to 3 Months and 5 Months
Description: Self-Efficacy will be assessed using the NIH PROMIS Self-Efficacy for Managing Daily Activities assessment. Minimum score = 0, Maximum score = 8. Higher numbers indicate greater self efficacy.
Time Frame: Baseline Visit, 3 months and 5 months
Population: as for outcome 1
Arm/Group | e Learning+Therapy (TEAACH)
Number analyzed (Participants) | 0

4. Secondary Outcome: Change in Social Isolation From Baseline to 3 Months and 5 Months
Description: Social Isolation will be assessed using the NIH PROMIS Social Isolation assessment. Minimum score = 0, Maximum score = 8. Higher numbers indicate less social isolation.
Time Frame: Baseline Visit, 3 months & 5 months
Population: as for outcome 1
Arm/Group | e Learning+Therapy (TEAACH)
Number analyzed (Participants) | 0

5. Secondary Outcome: Change in Emotional Support From Baseline to 3 Months and 5 Months
Description: Emotional Support will be assessed using the NIH PROMIS Emotional Support assessment. Minimum score = 0, Maximum score = 8. Higher numbers indicate greater emotional support.
Time Frame: Baseline Visit, 3 months (Post Treatment+/- 3 days), & 5 months (Follow up +/- 3 days)
Population: as for outcome 1
Arm/Group | e Learning+Therapy (TEAACH)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed
Description: The first subject was enrolled in August 2019 but study procedures could not begin until a cohort was enrolled as per study design. Hence, because of the covid shut down in March 2020 we did not enroll a complete cohort and the study stopped prior to beginning the group-related study procedures. Therefore, All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | e Learning+Therapy (TEAACH)
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-14): https://cdn.clinicaltrials.gov/large-docs/49/NCT04245449/Prot_SAP_000.pdf
  • Informed Consent Form (2019-08-14): https://cdn.clinicaltrials.gov/large-docs/49/NCT04245449/ICF_001.pdf